CLINICAL TRIAL: NCT05720182
Title: Validation of CPM#1 Compressibility in Healthy Volunteers in Rest and After Exercise
Brief Title: Non-invasive Measurement of Compartment Pressure: Reliability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kay van Heeswijk (Other)
Collaborators: CPM Sport AG Bern (Unknown)
Responsible Party: Sponsor-Investigator, Kay van Heeswijk, Coordinating Investigator, Maxima Medical Center
Organization: Maxima Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-MMC-098; NL.82601.015.22 (Other: CCMO)
Record Dates: First submitted 2023-01-18; First posted 2023-02-09 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: CEC Syndrome
Keywords: Non-invasive; Reliability; Healthy Volunteers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A performance validation pilot of the CPMX1 device in healthy volunteers. There will only be one study arm, no comparator, and no randomization.
Masking Description: No true masking possible, as the study only uses healthy participants and all participants will get measurements to both legs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy subjects are not subjected to any type of treatment besides non-invasive lower leg muscle compressibility measurements in rest and after exercise.
  All 35 healthy subjects will undergo four times four measurements in rest (m. tibialis anterior of both legs, using two different internal landmarks). These four times four measurements in rest will each be done by three observers.
  To measure the effect of exercise, compressibility will be measured immediately, one minute, and five minutes after a standard treadmill exercise at just one leg. The treadmill exercise and the corresponding measurements will be performed twice to address for measurements of both legs.
  Interventions: Device: Compremium Compressibility Measurement; Procedure: Treadmill Running; Other: Questionnaire

INTERVENTIONS:
Device: Compremium Compressibility Measurement — CPM#1 measurements:
  Step 1: Manual investigation to identify the compartment for compressibility measurements
  Step 2: Marking the location for compressibility measurements
  Step 3 - Examination with CPM#1
  * Place the probe on the target area
  * Identify correct landmark
  * Compress the compartment
  * Increase steadily the pressure applied by the CP probe to 80 mmHg.
Procedure: Treadmill Running — Exercise:
  Step 1: Participants will walk on a treadmill with standardized walking speed (5.0 km/hour) and slope (15%) for 5 minutes.
  Step 2: Immediate, one minute, and five minutes post-exercise CPM#1 measurements will be performed at one leg.
  Exercise and post-exercise CPM#1 measurements will be repeated for the other leg.
Other: Questionnaire — Questionnaires NIAPS questionnaire: Baseline NIAPS questionnaire with one additional question about leg dominance.
  Experience questionnaire: Scores 1-5, questioning the intensity, how painful, the nuisance, the duration of the study and the non-invasive pressure measurements.

SUMMARY:
The investigators want to investigate the reliability (variability) of a new device, that should be able to measure lower leg compartment pressure non-invasively. Therefore the tool is used under different circumstances. The introduced differences in circumstances are:

* Measurements at several time points
* Measurements using different anatomical landmarks
* Measurements by different researchers
* Measurements in rest and after exercise

This study's results are important to create a reliable measurement tools for patients with lower leg symptoms. In this way the diagnosis can be improved and as well the treatments given to the patients.

It is expected that the variability of the device will be low compared to current techniques.

DETAILED DESCRIPTION:
Chronic Exertional Compartment Syndrome (CECS) is one of the exercise-induced lower leg pathologies. Recognition by patients and physicians is not optimal. As a consequence, many patients are undiagnosed and are forced to stop their sporting activities. To diagnose CECS, a doctor should be alerted by a patient's history and a physical examination. If both suggestive of CECS, an invasive intra compartmental pressure measurement (ICPM) in the affected compartment may be performed. During the ICPM a catheter is placed into the muscle via a hollow needle. The ICPM is not flawless in terms of accuracy and reproducibility and has a low intra-observer reproducibility. Moreover, haematoma or other tissue damage may occur following an ICPM. Nevertheless, this invasive ICPM is in 2022 still considered the 'gold-standard' diagnostic tool for CECS, in the absence of a better one.

A novel non-invasive tool for CECS is possibly provided by measuring muscle tissue compressibility. The idea is, that muscle tissue with a high pressure (as in CECS patients) requires more external force to compress, compared to tissue with a low pressure. The study device used in this study, the CPM#1 device, is based on this principle. The CPM#1 device is non-invasive, not painful, very user friendly, and the measurement can be executed as an 'office procedure' in a couple of minutes. This study will focus on determining the reliability of the device in healthy volunteers.

The primary objective is

- To validate the inter-observer reliability of compressibility measurements with the CPM#1 device during rest in healthy volunteers.

Secondary objectives are

* To validate the intra-observer reliability of compressibility measurements with the CPM#1 device during rest in healthy volunteers.
* To investigate the effect of exercise on compressibility immediately, one minute, and five minutes after exercise in healthy volunteers.
* To map the invasiveness of the compressibility measurement with the CPM#1 device.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Healthy subjects will undergo several compressibility measurements, both before and after a treadmill exercise. They will also complete a NIAPS (Netwerk Inspannings Afhankelijke PijnSyndromen) questionnaire and an 'experience' questionnaire. The harm associated with the CPM#1 device is none. However, the subjects will not benefit from this study

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Proficient in speaking and reading Dutch

Exclusion Criteria:

* Presence of complaints suggestive of CECS, previously diagnosed with CECS or previous positive ICPM
* History of surgery or other trauma which penetrated the fascia of the leg
* Other concurrent limb pathologies or anomalies amongst others:
* Peripheral arterial or venous disease
* Muscle disorders, diabetes mellitus, peripheral neuropathies
* Unable to exercise for five minutes
* Open wound or painful bruise less than one week ago at site of measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Inter-class correlation | 1 session of approximately 90 minutes
  The primary endpoint of inter-observer variability will be the intraclass correlation coefficient (ICC) of agreement between three observers, four sites per subject, and four repetitions per measurement. The ICC will be assessed using a two-way random effects model. Both observers and subjects will be included as random effects. The first measurement for each location will be taken from every observer to calculate the ICC. Apart from that, the ICC will be measured using the average of the four repetitions of ratings, to estimate the effect on the ICC of repetitive measurements. "Good reliability" classification will be reached if the lower bound of the computed ICC confidence interval does not fall below 0.75.

SECONDARY OUTCOMES:
Intra-class correlation | 1 session of approximately 90 minutes
  The secondary endpoint of intra-observer variability will be the intraclass correlation coefficient (ICC) of agreement within three observers, four sites per subject, and four repetitions per measurement. The ICC will be assessed using a two-way random effects model. Both subjects and repetitions will be included as random effects. The repeated measures will be analysed for each observer separately and this agreement serves to address differences between observers. "Good reliability" classification will be reached if the lower bound of the computed ICC confidence interval does not fall below 0.75
Exercise effect on compressibility | Directly, 1 minute, and 5 minutes post-exercise
  The second secondary endpoint is the comparison between post-exercise (immediate, one minute, and five minutes) compressibility and rest compressibility. This will be analysed using a dependent sample t-test.
  Compressibility is expressed as a CP-value (defined as percentage reduction of the muscle length under two different types of pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Marc RM Scheltinga, Dr, Principal Investigator — Máxima Medisch Centrum
Locations (1):
- Máxima Medisch Centrum, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will only be used by the sponsor and anonymously with the subsiding party.

REFERENCES:
- [Background] Orlin JR, Lied IH, Stranden E, Irgens HU, Andersen JR. Prevalence of chronic compartment syndrome of the legs: Implications for clinical diagnostic criteria and therapy. Scand J Pain. 2016 Jul;12:7-12. doi: 10.1016/j.sjpain.2016.01.001. Epub 2016 Mar 4. PMID 28850498
- [Background] Maksymiak R, Ritchie E, Zimmermann W, Maliko N, van der Werve M, Verschure M, Hoencamp R. Historic cohort: outcome of chronic exertional compartment syndrome-suspected patients. BMJ Mil Health. 2021 Dec;167(6):387-392. doi: 10.1136/jramc-2019-001290. Epub 2020 Feb 3. PMID 32019808
- [Background] Vogels S, VAN Ark W, Janssen L, Scheltinga MRM. Fasciectomy for Recurrent Chronic Exertional Compartment Syndrome of the Anterior Leg. Med Sci Sports Exerc. 2021 Aug 1;53(8):1549-1554. doi: 10.1249/MSS.0000000000002631. PMID 33731658
- [Background] Houston A, Cosma G, Turner P, Bennett A. Predicting surgical outcomes for chronic exertional compartment syndrome using a machine learning framework with embedded trust by interrogation strategies. Sci Rep. 2021 Dec 20;11(1):24281. doi: 10.1038/s41598-021-03825-4. PMID 34931008
- [Background] Pedowitz RA, Hargens AR, Mubarak SJ, Gershuni DH. Modified criteria for the objective diagnosis of chronic compartment syndrome of the leg. Am J Sports Med. 1990 Jan-Feb;18(1):35-40. doi: 10.1177/036354659001800106. PMID 2301689
- [Background] Vogels S, Ritchie ED, Bakker EWP, Vogels MAJM, Zimmermann WO, Verhofstad MHJ, Hoencamp R. Measuring intracompartmental pressures for the chronic exertional compartment syndrome: Challenging commercially available devices and their respective accuracy. J Biomech. 2022 Apr;135:111026. doi: 10.1016/j.jbiomech.2022.111026. Epub 2022 Feb 28. PMID 35288313
- [Background] Large TM, Agel J, Holtzman DJ, Benirschke SK, Krieg JC. Interobserver Variability in the Measurement of Lower Leg Compartment Pressures. J Orthop Trauma. 2015 Jul;29(7):316-21. doi: 10.1097/BOT.0000000000000317. PMID 25756911
- [Background] Bloch A, Tomaschett C, Jakob SM, Schwinghammer A, Schmid T. Compression sonography for non-invasive measurement of lower leg compartment pressure in an animal model. Injury. 2018 Mar;49(3):532-537. doi: 10.1016/j.injury.2017.11.036. Epub 2017 Nov 27. PMID 29195681
- [Background] Herring MJ, Donohoe E, Marmor MT. A Novel Non-invasive Method for the Detection of Elevated Intra-compartmental Pressures of the Leg. J Vis Exp. 2019 May 31;(147). doi: 10.3791/59887. PMID 31205299
- [Background] Marmor MT, Barker JP, Matz J, Donohoe E, Herring MJ. A dual-sensor ultrasound based method for detecting elevated muscle compartment pressures: A prospective clinical pilot study. Injury. 2021 Aug;52(8):2166-2172. doi: 10.1016/j.injury.2021.02.054. Epub 2021 Feb 19. PMID 33640161
- [Background] Anwander H, Buchel L, Krause F, Siebenrock K, Schmid T. Tibial anterior compartment compressibility in healthy subject, measured using compression sonography. Injury. 2022 Feb;53(2):719-723. doi: 10.1016/j.injury.2021.12.014. Epub 2021 Dec 17. PMID 34963511
- See also: Sealed Envelope LTD. Create a blocked randomisation list — https://www.sealedenvelope.com/
- See also: Winkes MB, Bloo H, Hoogeveen AR, Scheltinga M. Het chronisch inspanningsgebonden compartimentsyndroom van het onderbeen. Physios. 2018;4:9. — https://www.physios.nl/artikelen/artikel/t/het-chronisch-inspanningsgebonden-compartimentsyndroom-van-het-onderbeen
- See also: Meehan WP, O'Brien MJ. Chronic exertional compartment syndrome UpToDate: UpToDate; 2020 — https://www.uptodate.com/contents/chronic-exertional-compartment-syndrome

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT05720182/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT05720182/ICF_001.pdf